CLINICAL TRIAL: NCT00174798
Title: A Randomized, Double-blind, Placebo and Active-controlled Efficacy and Safety Study of SSR240600C in Patients With Overactive Bladder (OAB) or Urge Urinary Incontinence (UUI)
Brief Title: MILADY: A Randomized, Placebo-controlled Safety and Efficacy Trial of SSR240600C in Treatment of Overactive Bladder or Urge Urinary Incontinence.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ACT5190; SSR240600C
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2012-02-02 (Estimated); Status verified 2012-02

CONDITIONS: Overactive Bladder
Keywords: Cystometry NK1 Antagonist SSR240600C
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Tolterodine Tartrate

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- SSR240600C (Experimental)
  Interventions: Drug: SSR240600C
- Tolterodine (Active Comparator)
  Interventions: Drug: Tolterodine

INTERVENTIONS:
Drug: SSR240600C — once daily
  Arms: SSR240600C
Drug: Placebo — oral
  Arms: Placebo
Drug: Tolterodine — once daily
  Arms: Tolterodine

SUMMARY:
To evaluate the safety and efficacy of SSR240600C versus placebo on clinical and cystometric parameters in patients with OAB and UUI.

DETAILED DESCRIPTION:
Prospective, randomized, parallel group, double-dummy, placebo and active-controlled (Detrol LA - tolterodine) trial wherein patients with OAB or UUI will receive single daily does of either SSR240600C 500 mg, tolterodine 4 mg or placebo for four weeks. Baseline and end of study cystometry will be performed; daily symptom diaries will be completed during the trial and health-related quality of life will be measured before and after study drug treatment. Patients will be followed-up one week after completion of the trial. Study participation will include 5 visits over a period of six weeks.

ELIGIBILITY:
Inclusion Criteria:

* Females between 18 and 75 years, inclusive Clinical diagnosis of OAB/UUI (symptoms of frequent micturition, urinary urgency)
* Bladder capacity </= 300 mL by cystometry

Exclusion Criteria:

* History of interstitial cystitis, bladder outlet obstruction or other significant genitourinary disorder
* Current urinary tract infection
* Neurological bladder dysfunction
* Treatment with drugs that may interfere with CYP3A4 metabolic function
* History of stress urinary incontinence

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2005-05; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Change in bladder capacity as determined by cystometric parameters from baseline to end of treatment.

SECONDARY OUTCOMES:
Change from baseline to end of treatment in:maximum detrusor pressure,volume ar first desire to void,volume at first unstable contraction,micturition frequence,urgency episodes,nocturia episodes,incontinence episodes,HRQOL and overall improvement

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (22):
- United States (22):
  - Hope Research LLC, Phoenix, Arizona
  - Research Tuscon, Tuscon, Arizona
  - Medical Center for Clinical Research, San Diego, California
  - Genitourinary Surgical Consultants, Denver, Colorado
  - Connecticut Clinical Research Center, Urology Specialists, Waterbury, Connecticut
  - Miami Research Associates, Miami, Florida
  - Southeastern Research Group, Tallahassee, Florida
  - Atlanta Women's Research Institute, Alpharetta, Georgia
  - Mount Vernon Clinical Research, Atlanta, Georgia
  - Soapstone Center for Education & Clinical Research, Decatur, Georgia
  - Urology of Indiana, Greenwood, Indiana
  - Metropolitan Urology, Jeffersonville, Indiana
  - Rockhill Medical Plaza, Kansas City, Missouri
  - Hudson Valley Urology Center, Kingston, New York
  - Hudson Valley Urology, Poughkeepsie, New York
  - Daniel Laury, Medford, Oregon
  - Philadelphia Women's Research, Philadelphia, Pennsylvania
  - Clinical Trials Research Services, Pittsburgh, Pennsylvania
  - University Urological Research Institute, Providence, Rhode Island
  - Advanced Research Associates, Corpus Christi, Texas
  - Tacoma Women's Specialists Research, Tacoma, Washington
  - Midwest Research SpecialistsSt. Michael's Hospital, Milwaukee, Wisconsin